CLINICAL TRIAL: NCT02856399
Title: Long-term Effects of Methadone for Cancer Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0523
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Cancer Pain
Keywords: methadone; cancer pain; long term effect
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The methadone is an useful opioid for the cancer pain treatment, mostly used in second or last line during the opioid rotation. The Methadone had an anti-MNDA effect, and clinicians agree that the methadone could have an effect in neuropathic cancer pain. During a previous study the investigators find that the pain was still improving after the week 2, but they had only a small number of patients still included at this stage and they cannot conclude.

The investigators decide to follow up systematically all the patients undergoing a methadone treatment for cancer pain, at day 28, to study the hypothesis about the long-term pain improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with t methadone for cancer pain in opioid rotation
* Able to fill the questionnaire
* Performance status (PS) from 0 to 2

Exclusion Criteria:

* Patients PS 3
* Unable to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a methadone treatment for cancer pain
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Difference between EVA pain score at Day 28 and Day 0 | pain score measure at Day 0 and Day 28
  long-term effects of methadone for cancer pain

SECONDARY OUTCOMES:
Change in score of neuropathic pain intensity NPSI | Day 0 and Day 28
Change in depression and anxiety score HADS | Day 0 and Day 28
Change in quality of life score QOL C30 | Day 0 and Day 28
Side effect record | up to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Marilene FILBET, Pr Associate, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Unité de Soins Palliatifs - Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, 165 Chemin du Grand Revoyet, Pierre-Bénite, France